CLINICAL TRIAL: NCT01266980
Title: An Open-label, Non-randomized Pharmacokinetic and Safety Study of Repeat Doses of Fluticasone Furoate and GW642444M Combination in Healthy Subjects and in Subjects With Severe Renal Impairment.
Brief Title: A Study to Assess the Effects of Repeat Doses of Fluticasone Furoate and GW642444M Combination in Healthy Subjects and in Subjects With Severe Impairment.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 113970
Record Dates: First submitted 2010-12-23; First posted 2010-12-24 (Estimated); Last update posted 2017-08-03 (Actual); Status verified 2017-08

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: cortisol; renal impairment; serum potassium; pharmacokinetics; Fluticasone furoate; heart rate
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Severe Renal Imparement (Experimental): Nine subjects with severe renal impairment (as defined by a Clcr<30mL/min) will be recruited for this study. they will receive FF/ GW642444M (200/25mcg) once daily for 7 days.
  Interventions: Drug: Inhaled FF/ GW642444M (200/25mcg)
- Matched healthy volunteers (Experimental): For each of the 9 renally impaired subjects a healthy control subject (as defined by a Clcr>80mL/min matched to the severe subjects based on gender, ethnicity, body mass index (±15%) and age (±5 years)) will be recuited. They will receive FF/ GW642444M (200/25mcg) once daily for 7 days.
  Interventions: Drug: Inhaled FF/ GW642444M (200/25mcg)

INTERVENTIONS:
Drug: Inhaled FF/ GW642444M (200/25mcg) — All subjects will be assigned to take FF/ GW642444M (200/25mcg) combination once daily for 7 days.

SUMMARY:
This study will assess the saftey of giving fluticasone furoate 200mcg/GW642444M 25mcg once daily for 7 days to patients with severe renal imparement. The results of this study will aid in deciding whether a FF/GW642444M doseadjustment is justified in subjects with severe renal impairment and in estimating any such adjustments.

DETAILED DESCRIPTION:
This is an open-label, non-randomized study which will assess the pharmacokinetics and safety following 7 days once daily dose of inhaled FF/ GW642444M (200/25mcg) in subjects with renal impairment. Nine subjects with severe renal impairment (as defined by a Clcr<30mL/min) will be recruited along with healthy control subjects (as defined by a Clcr>80mL/min matched to the severe subjects based on gender, ethnicity, body mass index (±15%) and age (±5 years)). All subjects will receive fluticasone furoate 200mcg/GW642444M 25mcg once daily for 7 days. The results of this study will aid in deciding whether a FF/GW642444M dose adjustment is justified in subjects with severe renal impairment and in estimating any such adjustments.

ELIGIBILITY:
Inclusion Criteria:

A subject will be eligible for inclusion in this study only if all of the following criteria apply:

1. Male or female between 18 and 70 years of age inclusive, at the time of signing the informed consent.
2. A female subject is eligible to participate if she is of:

   * Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 MlU/ml and estradiol < 40 pg/ml (<140 pmol/L) (healthy subjects only) is confirmatory]. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the contraception methods in Section 8.1 if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrollment. For most forms of HRT, at least 2-4 weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method.
   * Child-bearing potential and agrees to use one of the contraception methods listed in Section 8.1 for an appropriate period of time (as determined by the product label or investigator) prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to use contraception until completion of the follow-up visit.
3. BMI within the range 19.0 - 33.0 kg/m^2 (inclusive).
4. Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
5. Single QTcF < 450 msec; or QTcF < 480 msec in subjects with Bundle Branch Block.
6. Able to satisfactorily use the dry powder inhaler.

   Healthy Subjects:
7. Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures or outcome.
8. AST, ALT, alkaline phosphatase and bilirubin ≤ 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
9. Creatinine clearance > 80mL/min calculated by the Cockcroft-Gault equation using serum creatinine.

   Renally Impaired Subjects:
10. AST and ALT < 2xULN; alkaline phosphatase and bilirubin ≤ 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
11. Creatinine clearance < 30mL/min calculated by the Cockcroft-Gault equation using serum creatinine.
12. Subjects with renal insufficiency must have stable renal function defined as ≤ 25% difference in creatinine clearance assessed on two occasions. Renal function will be based on estimated creatinine clearance (CLcr) calculated by the Cockcroft-Gault equation using serum creatinine obtained on two occasions separated by at least 4 weeks within the last 3 months (historic data is permitted for the first measurement).

Exclusion Criteria:

A subject will not be eligible for inclusion in this study if any of the following criteria apply:

1. Suffered a lower respiratory tract infection in the 4 weeks before the screening visit.
2. Taken oral corticosteroids less than 8 weeks before the screening visit.
3. Taken inhaled, intranasal or topical steroids less than 4 weeks before the screening visit.
4. Any subject with either documented cirrhosis or a history consistent with a diagnosis of cirrhosis.
5. A positive pre-study drug/alcohol screen.
6. A positive test for HIV antibody.
7. The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
8. Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
9. Use of nephrotoxic medications 4 weeks before dosing.
10. Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
11. Pregnant females as determined by positive serum or urine hCG test at screening or prior to dosing.
12. Lactating females.
13. The subject has been treated for or diagnosed with depression within six months of screening or has a history of significant psychiatric illness.
14. Unwillingness or inability to follow the procedures outlined in the protocol.
15. Subject is mentally or legally incapacitated.
16. History of sensitivity to heparin or heparin-induced thrombocytopenia.
17. Subjects with smoking history of >10 cigarettes per day or regular use of tobacco- or nicotine-containing products, within 6 months prior to screening.
18. History of severe milk protein allergy.
19. Any adverse reaction including immediate or delayed hypersensitivity to any beta2- agonist, sympathomimetic drug, or any intranasal, inhaled, or systemic corticosteroid therapy. Known or suspected sensitivity to the constituents of the Novel DPI (i.e., lactose or magnesium stearate). History of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
20. Consumption of red wine, seville oranges, grapefruit or grapefruit juice and/or pummelos, exotic citrus fruits, grapefruit hybrids or fruit juices from 7 days prior to the first dose of study medication.

    Healthy Subjects:
21. If, in the opinion of the examining physician, an unstable cardiovascular, renal, hepatic, pulmonary, endocrine, metabolic, neurological, haematological or gastrointestinal condition is present or any other medical condition which the investigator considers sufficiently serious to interfere with the conduct, completion, or results of this trial or constitutes an unacceptable risk to the subject.
22. Subjects with any predisposing condition that might interfere with the absorption, distribution, metabolism or excretion of drugs or any previous gastrointestinal (GI) surgery (except appendectomy or cholecystectomy more than three months prior to the study) or condition (including pancreatitis or acute cholecystitis) which the investigator considers sufficiently significant to interfere with the conduct, completion, or results of this trial or constitutes an unacceptable risk to the subject.
23. Urinary tract or bladder infection within 4 weeks of the first scheduled administration of study drug.
24. A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
25. Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
26. History of regular alcohol consumption within 6 months of the study defined as:

    • An average weekly intake of >21 units for males or >14 units for females. One unit is equivalent to 8 g of alcohol: a half-pint (~240 ml) of beer, 1 glass (125 ml) of wine or 1 (25 ml) measure of spirits.
27. Hemoglobin or hematocrit below the reference range at screening.
28. Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inhibitor) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.

    Renally Impaired Subjects:
29. Life expectancy less than 3 months.
30. Hemoglobin less than 8.5 g/dL.
31. Subjects on hemodialysis treatment.
32. Subjects who, within the past six months, have had a history of significant drug abuse or alcohol abuse.
33. Subjects who need to take any concomitant medication, either prescribed or overthe- counter, which may in the opinion of the Investigator, interfere in any way with the study procedure or be a safety concern (see Section 9 for the list of permitted concurrent medications). In particular subjects taking medications that significantly inhibit P450 CYP3A4 (e.g. ketaconazole) must not be included in this study.
34. If in the opinion of an examining physician an unstable cardiovascular, pulmonary or hepatic condition is present, or any other medical condition which the investigator considers sufficiently serious to interfere with the conduct, completion, or results of this trial or constitutes an unacceptable risk to the subject.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2010-11-18 (Actual); Primary Completion 2011-03-22 (Actual); Study Completion 2011-03-22 (Actual)

PRIMARY OUTCOMES:
Fluticasone furoate and GW642444 pharmacokinetics (AUC(0-t), AUC (0-8),Cmax, tmax,) on Day 1 and 7 and AUC(0-24) and t½ on Day 7. | 1 Month

SECONDARY OUTCOMES:
Serum cortisol weighted mean over 24 hours on Days -1 and 7 | 1 Month
Maximum heart rate over time period 0-4 hours on Day 7. | 1 Month
Minimum serum potassium values over time period 0-4 hours on Day 7. | 1 Month
General safety and tolerability endpoints: adverse events, blood pressure, heart rate, 12-lead ECG, clinical laboratory safety tests. | 1 Month

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Prague, Czechia

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Allen A, Davis A, Hardes K, Tombs L, Kempsford R. Influence of renal and hepatic impairment on the pharmacokinetic and pharmacodynamic properties and tolerability of fluticasone furoate and vilanterol in combination. Clin Ther. 2012 Dec;34(12):2316-32. doi: 10.1016/j.clinthera.2012.11.001. Epub 2012 Nov 30. PMID 23200625
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 113970 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/113970?search=study&study_ids=113970#rs
- Available data/document: Individual Participant Data Set: 113970 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 113970 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 113970 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 113970 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 113970 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 113970 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 113970 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register